CLINICAL TRIAL: NCT00807118
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 2-Cohort, 3-Way Crossover Study To Determine Bioequivalence Of 4 Mg And 8 Mg Fesoterodine SR Tablet Of Commercial Formulation And 8 Mg Fesoterodine SR Tablet Between Formulation E(1) And Formulation F And Investigate Food Effect On Commercial Formulation In Healthy Subjects.
Brief Title: Phase 1, Single Dose, Crossover Study to Determine Bioequivalence and to Investigate Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0221052
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Therapeutic Equivalency; Food
Keywords: bioequivalence, food effect
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Cohort I) (Experimental)
  Interventions: Drug: Fesoterodine
- B (Cohort I) (Experimental)
  Interventions: Drug: Fesoterodine
- C (Cohort I) (Experimental)
  Interventions: Drug: Fesoterodine
- B (Cohort II) (Experimental)
  Interventions: Drug: Fesoterodine
- D (Cohort II) (Experimental)
  Interventions: Drug: Fesoterodine
- E (Cohort II) (Experimental)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Single dose of 2 x 4 mg tab in formulation F under fed condition
  Arms: A (Cohort I)
Drug: Fesoterodine — Single dose of 1 x 8 mg tab in formulation F under fed condition
  Arms: B (Cohort I)
Drug: Fesoterodine — Single dose of 1 x 8 mg tab in formulation E(1) under fed condition
  Arms: C (Cohort I)
Drug: Fesoterodine — Single dose of 1 x 8 mg tab in formulation F under fed condition
  Arms: B (Cohort II)
Drug: Fesoterodine — Single dose of 2 x 4 mg tab in formulation F under fasted condition
  Arms: D (Cohort II)
Drug: Fesoterodine — Single dose of 1 x 8 mg tab in formulation F under fasted condition
  Arms: E (Cohort II)

SUMMARY:
Primary objectives are to demonstrate bioequivalence between 4 and 8 mg of commercial formulation in both under fasted and fed condition, and bioequivalence between formulation E(1) used in Japanese pivotal study and commercial formulation in 8 mg. Secondary objective is to assess food effect on 8 mg tablet of commercial formulation. These objectives are set to get data for Japanese regulatory submission.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subject

Exclusion Criteria:

* Evidence or history of clinically significant findings at screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
AUCt and Cmax of 5-HMT after single oral administration of 2 tabs of 4 mg fesoterodine SR tablets of formulation F and 1 tab of 8 mg fesoterodine SR tablets of formulation F under fed condition | Day 1 and 2
AUCt and Cmax of 5-HMT after single oral administration of 2 tabs of 4 mg fesoterodine SR tablets of formulation Fand 1 tab of 8 mg fesoterodine SR tablets of formulation F under fasted condition | Day 1 and 2
AUCt and Cmax of 5-HMT under after single oral administration of 1 tab of 8 mg fesoterodine SR tablets of formulation F and 1 tab of 8 mg fesoterodine SR tablet of formulation E(1) | Day 1 and 2

SECONDARY OUTCOMES:
Tmax, AUClast, AUCinf, kel, t1/2 and MRT of all treatment | Day 1 and 2
AUCt and Cmax after single oral administration of 8 mg fesoterodine SR tablets of formulation F under fed condition in cohort II | Day 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221052&StudyName=Phase%201%2C%20single%20dose%2C%20crossover%20study%20to%20determine%20bioequivalence%20and%20to%20investigate%20food%20effect